CLINICAL TRIAL: NCT00748306
Title: A Randomised, Double-blind, Placebo-controlled, 2-period Cross-over Study to Evaluate the Effect of Treatment With GSK2190915 on the Allergen-induced Asthmatic Response in Subjects With Mild Asthma
Brief Title: Study in Mild Asthmatic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 111834
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
Keywords: challenge; early asthmatic response; mild asthmatics; Allergen; methacholine
MeSH Terms: conditions — Asthma | interventions — 3-(3-tert-butylsulfanyl-1-(4-(6-ethoxypyridin-3-yl)benzyl)-5-(5-methylpyridin-2-ylmethoxy)-1H-indol-2-yl)-2,2-dimethylpropionic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK2190915 (Experimental): Intervention
  Interventions: Drug: GSK2190915 - 100mcg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2190915 - 100mcg — GSK2190915 is a high affinity 5-lipoxygenase-activating protein (FLAP) inhibitor
  Other Names: GSK2190915
  Arms: GSK2190915
Drug: Placebo — Matching Intervention Drug
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and usefulness of GSK2190915 in asthmatic patients who develop asthma symptoms following being challenged.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 to 55 years inclusive.
2. Body mass index within the range 18.5-35.0 kilograms/metre2 (kg/m2).
3. Female subjects must be of non childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 40 pg/ml (<140 pmol/L) or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
4. Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 5 terminal half-live post-last dose.
5. Documented history of bronchial asthma, first diagnosed at least 6 months prior to the screening visit and currently being treated only with intermittent short-acting beta -agonist therapy by inhalation.
6. Pre-bronchodilator FEV1 >70% of predicted at screening.
7. Sensitivity to methacholine with a provocative concentration of methacholine resulting in a 20% fall in FEV1 (PC20 methacholine) of <8 mg/mL at screening
8. Subjects who are able to produce acceptable induced sputum samples (as defined in the Study procedures Manual).
9. Subjects who are current non-smokers who have not used any tobacco products in the 6-month period preceding the screening visit and have a pack history of ≤10 pack years.

   [number of pack years = (number of cigarettes per day/20) x number of years smoked]
10. Demonstration of a positive wheal and flare reaction (≥3 mm relative to negative control) to at least one allergen from a battery of allergens (including house dust mite, grass pollen and cat hair) on skin prick testing at screening, or within 12 months of study start.
11. Screening allergen challenge demonstrates that the subject experiences both an early and late asthmatic response. The early asthmatic response must include a fall in FEV1 of ≥20% from the post saline value, on at least one occasion, between 5 and 30 minutes after the final concentration of allergen. The late asthmatic response must include a fall in FEV1 of ≥ 15% from the post saline value, on at least three occasions, two of which must be consecutive, between 4 and 10 hours after the final concentration of allergen.
12. Signed and dated written informed consent is obtained from the subject
13. The subject is able to understand and comply with the protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Past or present disease, which as judged by the investigator or medical monitor, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, gastrointestinal disease, hepatic disease, renal disease, haematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to chronic bronchitis, emphysema, bronchiectasis or pulmonary fibrosis).
2. Clinically significant abnormalities in safety laboratory analysis at screening.
3. Subject has known history of hypertension or is hypertensive at screening. Hypertension at screening is defined as persistent systolic BP >150 mmHg or diastolic BP > 90mmHg.
4. Respiratory tract infection and/or exacerbation of asthma within 4 weeks prior to the first dose of study medication.
5. History of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest and/or hypoxic seizures.
6. Symptomatic with hay fever at screening or predicted to have symptomatic hayfever during the time of study.
7. Administration of oral or injectable steroids within 5 weeks of screening or intranasal and/or inhaled steroids within 4 weeks of the screening visit.
8. Unable to abstain from other medications including non-steroidal anti-inflammatory drugs (NSAIDs), anti-depressant drugs, anti-histamines and anti-asthma, anti-rhinitis or hay fever medication, other than short acting inhaled beta-agonists and paracetamol (up to 4 g per day) for the treatment of minor ailments eg headache from 14 days before screening until the follow-up visit.
9. Unable to abstain from short acting beta agonists as described in the restrictions section.
10. If, after 2 concurrent administrations of saline during the allergen challenge at screening the subjects still have a fall in FEV1 of greater than 10%.
11. The subject has participated in a study with a new molecular entity during the previous 3 months or has participated in 4 or more clinical studies in the previous 12 months prior to the first dosing day.
12. History of being unable to tolerate or complete methacholine and/or allergen challenge tests.
13. Subject is undergoing allergen desensitisation therapy.
14. There is a risk of non-compliance with study procedures.
15. History of blood donation (500 mL) within 3 months of starting the clinical study.
16. The subject regularly drinks more than 28 units of alcohol in a week if male, or 21 units per week if female. One unit of alcohol is defined as a medium (125 ml) glass of wine, half a pint (250 ml) of beer or one measure (25 ml) of spirits.
17. The subject has a screening QTc value of >450msec, PR interval outside the range 120 to 220msec or an ECG that is not suitable for QT measurements (e.g. poorly defined termination of the T-wave).
18. The subject has tested positive for hepatitis C antibody or hepatitis B surface antigen.
19. The subject has tested positive for HIV antibodies.
20. The subject has a positive pre-study urine cotinine/ breath carbon monoxide test or urine drug or urine or breath alcohol screen. A minimum list of drugs that will be screened for include Amphetamines, Barbiturates, Cocaine, Opiates, Cannabinoids and Benzodiazepines.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2008-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change in FEV1% from 0-2 hrs | 0-2 hours

SECONDARY OUTCOMES:
Late Asthmatic Response (LAR): minimum FEV1 and weighted mean FEV1 between 4-10 hours after allergen challenge on Day 3 of each treatment period. | 4 - 10 hours after allergen challenge
Incidence of treatment emergent adverse events. | Duration of Study
Vital signs, ECG, FEV1, Biomarkers(LTE4, LTB4 and IgE) and safety laboratory parameters. | Duration of Study
Assessment of FEV1 post-dose on Days 1, 3, (post-dose on Days 3 prior to allergen challenge) and Day 6 of each treatment period. | upto Day 3
Concentration of exhaled nitric oxide post-dose on Day 3, 4 and 6 of each treatment period. | Day 3 - 6
Provocative concentration of methacholine resulting in a 20% reduction in FEV1 (PC20) on Day 4 of each treatment period. | Day 4
Biomarkers (LTE4, LTB4 and IgE) of inflammation in blood, urine and sputum of each treatment period.
Assessment of established markers of anti-inflammatory activity in sputum on Day 4 and Day 6. | Day 4
Derived appropriate PK parameters for GSK2190915. | Duration of Study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Leiden, Netherlands
- United Kingdom (2):
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kent SE, Boyce M, Diamant Z, Singh D, O'Connor BJ, Saggu PS, Norris V. The 5-lipoxygenase-activating protein inhibitor, GSK2190915, attenuates the early and late responses to inhaled allergen in mild asthma. Clin Exp Allergy. 2013 Feb;43(2):177-86. doi: 10.1111/cea.12002. PMID 23331559
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 111834 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111834 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111834 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111834 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111834 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111834 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111834 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register